CLINICAL TRIAL: NCT06431243
Title: An Open, Multicenter Phase Ib/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of the Purinostat Mesylate for Injection in Combination Therapy for Advanced Solid Tumors
Brief Title: A Clinical Study of Purinostat Mesylate for Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZLPM-003-1.0
Record Dates: First submitted 2024-05-20; First posted 2024-05-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A0 group (Experimental): Cohort A0 is for patients with locally advanced or metastatic breast cancer treated with PM. The cohort doses are escalated in the order of 11.2 mg/m2, 15.0 mg/m2, and XX mg/m2 (if the SMC assesses that there are safety risks in the monotherapy escalation starting dose group, it can be reduced to 8.4 mg/m2 or a dose determined by the SMC). In Cohort A0, subjects in the dose-escalation group all receive PM intravenous infusion on days 1, 4, 15, and 18 of each cycle, with a 28-day cycle (within the same dosing cycle, the interval between two doses is at least ≥48 h), and the maximum duration of dosing does not exceed 96 weeks.
  Interventions: Drug: A0/B0 group Purinostat Mesylate 11.2mg/m2; Drug: A0/B0 group Purinostat Mesylate 15mg/m2
- A group (Experimental): Cohort A is for patients with HR+/HER2- (hormone receptor positive/human epidermal growth factor receptor 2 negative) advanced breast cancer treated with PM in combination with fulvestrant. In Cohort A, subjects in the dose-escalation group all receive PM intravenous infusion on days 1, 4, 15, and 18 of each cycle, with a 28-day cycle (within the same dosing cycle, the interval between two doses is at least ≥48 h); fulvestrant (FS) is administered as two 5 mL injections slowly into the buttocks on days 1 and 15 of the first cycle, with one injection per buttock (1-2 minutes/5 mL), and starting from the second cycle, 500 mg (specification 5 mL: 0.25 g) is given once on the first day of each cycle (CnD1), with a 28-day cycle. Based on the results obtained in the dose-escalation phase, the necessity of the Phase IIa expansion cohort and the dosing of PM will be determined by the SMC after discussion.
  Interventions: Drug: A group Purinostat Mesylate 6mg/m2; Drug: A group Purinostat Mesylate 8.4mg/m2; Drug: A group Purinostat Mesylate 11.2mg/m2; Drug: A group Purinostat Mesylate 15 mg/m2
- B0 group (Experimental): Cohort B0 is for patients with advanced solid tumors treated with PM. The cohort doses are escalated in the order of 11.2 mg/m2, 15.0 mg/m2, and XX mg/m2 (if the SMC assesses that there are safety risks in the monotherapy escalation starting dose group, it can be reduced to 8.4 mg/m2 or a dose determined by the SMC). In Cohort B0, subjects in the dose-escalation group all receive PM intravenous infusion, with a dosing frequency of BiW (twice weekly), for continuous dosing over 2 weeks, that is, on days 1, 4, 8, and 11 of each cycle, with a 21-day cycle (within the same dosing cycle, the interval between two doses is at least ≥48 h), and the maximum duration of dosing does not exceed 96 weeks.
  Interventions: Drug: A0/B0 group Purinostat Mesylate 11.2mg/m2; Drug: A0/B0 group Purinostat Mesylate 15mg/m2
- B group (Experimental): Cohort B is for patients with advanced solid tumors treated with PM in combination with tislelizumab. In Cohort B, subjects in the dose-escalation group all receive PM intravenous infusion on days 1, 4, and 8 of each cycle, with a 21-day cycle (within the same dosing cycle, the interval between two doses is at least ≥48 h). Tislelizumab is administered as a 200 mg intravenous infusion, once every 3 weeks, on the first day of each cycle. Based on the results obtained in the dose-escalation phase, the necessity of the Phase IIa expansion cohort and the dosing will be determined by the Safety Monitoring Committee (SMC) after discussion.
  Interventions: Drug: B group Purinostat Mesylate 6 mg/m2; Drug: B group Purinostat Mesylate 8.4 mg/m2; Drug: B group Purinostat Mesylate 11.2mg/m2; Drug: B group Purinostat Mesylate 15mg/m2

INTERVENTIONS:
Drug: A0/B0 group Purinostat Mesylate 11.2mg/m2 — Purinostat Mesylate 11.2mg/m2
  Arms: A0 group; B0 group
Drug: A0/B0 group Purinostat Mesylate 15mg/m2 — Purinostat Mesylate 15mg/m2
  Arms: A0 group; B0 group
Drug: A group Purinostat Mesylate 6mg/m2 — Purinostat Mesylate 6mg/m2 + FS 500mg
  Arms: A group
Drug: A group Purinostat Mesylate 8.4mg/m2 — Purinostat Mesylate 8.4mg/m2 + FS 500mg
  Arms: A group
Drug: A group Purinostat Mesylate 11.2mg/m2 — Purinostat Mesylate 11.2mg/m2 + FS 500mg
  Arms: A group
Drug: A group Purinostat Mesylate 15 mg/m2 — Purinostat Mesylate 15 mg/m2 + FS 500mg
  Arms: A group
Drug: B group Purinostat Mesylate 6 mg/m2 — Purinostat Mesylate 6mg/m2 + Tislelizumab 200mg
  Arms: B group
Drug: B group Purinostat Mesylate 8.4 mg/m2 — Purinostat Mesylate 8.4mg/m2 + Tislelizumab 200mg
  Arms: B group
Drug: B group Purinostat Mesylate 11.2mg/m2 — Purinostat Mesylate 11.2mg/m2 + Tislelizumab 200mg
  Arms: B group
Drug: B group Purinostat Mesylate 15mg/m2 — Purinostat Mesylate 15mg/m2 + Tislelizumab 200mg
  Arms: B group

SUMMARY:
Primary Objectives Phase Ib To evaluate the safety and tolerability of Purinostat Mesylate in combination therapy for advanced solid tumors; and to explore the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of Purinostat Mesylate in combination therapy in patients with advanced solid tumors.

To determine the recommended Phase II dose (RP2D) of Purinostat Mesylate in combination therapy for advanced solid tumors.

Phase IIa To further evaluate the preliminary efficacy of Purinostat Mesylate in combination therapy in patients with advanced solid tumors.

Secondary Objectives Phase Ib To evaluate the safety and tolerability of Purinostat Mesylate Monotherapy for the treatment of advanced solid tumors; To evaluate the preliminary efficacy of Purinostat Mesylate in combination therapy in patients with advanced solid tumors; To evaluate the pharmacokinetic characteristics of Purinostat Mesylate in combination therapy for the treatment of advanced solid tumors.

Phase IIa To further evaluate the safety and tolerability of Purinostat Mesylate in combination therapy for advanced solid tumors.

To evaluate the pharmacokinetic characteristics of Purinostat Mesylate in combination therapy for advanced solid tumors.

Exploratory Objectives To assess the pharmacodynamic characteristics in Purinostat Mesylate combination therapy for advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria:

1. Age: ≥18 years and ≤75 years, regardless of gender.
2. At least one measurable lesion as defined by RECIST 1.1 during the screening period (for the breast cancer cohort in the dose-escalation phase, measurable lesions are not required if the participant has only bone metastases).
3. Phase Ib:

Monotherapy Dose-Escalation Phase:

1. Monotherapy in Cohort A0 (Breast Cancer):

   Histologically or cytologically confirmed locally advanced or metastatic breast cancer that has failed standard treatment, for which no standard treatment is available, or for which standard treatment is not suitable at the current stage.
2. Monotherapy in Cohort B0 (Solid Tumors):

Histologically or cytologically confirmed locally advanced or metastatic solid tumors that have failed standard treatment, for which no standard treatment is available, or for which standard treatment is not suitable at the current stage. This includes but is not limited to triple-negative breast cancer, colorectal cancer, and urothelial cancer.

Combination Therapy Dose-Escalation Phase:

1. Combination with Fulvestrant in Cohort A (Breast Cancer):

   * Histologically or cytologically confirmed breast cancer in perimenopausal, premenopausal, or postmenopausal women with estrogen receptor (ER)-positive, progesterone receptor (PgR)-negative or positive, and non-HER2-positive (including HER2-negative and low-expression) disease.
   * Participants must have progressed or recurred after at least one line of endocrine therapy (regardless of whether it was in the advanced, metastatic, or neoadjuvant chemotherapy setting), with up to two lines of prior chemotherapy allowed.
   * Ineligible for surgical resection.
   * Definition of menopause must meet one of the following criteria:

     1. Previous bilateral oophorectomy;
     2. Age 60 years or older;
     3. Under 60 years old, with no chemotherapy, tamoxifen, toremifene, or ovarian suppression therapy within the past year, and naturally postmenopausal for more than 12 months with serum follicle-stimulating hormone and estradiol levels in the postmenopausal range;
     4. Under 60 years old, currently receiving tamoxifen or toremifene therapy, with serum follicle-stimulating hormone and estradiol levels within the postmenopausal range on two consecutive tests;
     5. If the above criteria are not met, the participant is considered premenopausal or perimenopausal. Female participants must meet the following criteria: Initiation of luteinizing hormone-releasing hormone (LHRH) agonists such as goserelin or leuprorelin at least 28±2 days before the first dose of study drug (participants who have already been using LHRH agonists for ≥21 days and <26 days before the first dose must have hormone levels meeting the criteria), and continued use of such drugs throughout the study treatment period.
2. Combination with Tislelizumab in Cohort B (Solid Tumors):

   * Histologically or cytologically confirmed locally advanced or metastatic solid tumors that have failed standard treatment, for which no standard treatment is available, or for which standard treatment is not suitable at the current stage.
   * The definition of failure of standard treatment for each tumor type is as follows:

     1. Non-small cell lung cancer: Metastatic patients without driver gene mutations: Progression or recurrence after at least second-line treatment (including platinum-based chemotherapy); Patients with tumors harboring EGFR, ROS1, ALK, or other driver gene mutations should have experienced failure of targeted therapy for these mutations and then progressed or recurred after at least second-line treatment (including platinum-based chemotherapy).
     2. Small cell lung cancer: Progression or recurrence after at least second-line treatment.
     3. Colorectal cancer: Progression or recurrence after at least second-line treatment (standard chemotherapy regimens previously received include fluorouracil or its derivatives, oxaliplatin, and irinotecan. Patients with BRAF V600E mutation should have received BRAF inhibitors. Patients with MSIH/dMMR should have received PD-1/PD-L1 therapy).
     4. Head and neck squamous cell carcinoma: Progression or recurrence after at least second-line treatment (including platinum-based chemotherapy).
     5. Urothelial cancer: Progression or recurrence after at least second-line treatment (recommended treatment regimens include PD-1/PD-L1 therapy, platinum-based chemotherapy, taxane chemotherapy, Disitamab Vedotin, and vinflunine. Patients with FGFR2/3 mutations should have received erdafitinib).
     6. Esophageal cancer: Progression or recurrence after at least second-line treatment (including platinum-based chemotherapy).
     7. Cervical cancer: Progression or recurrence after at least second-line treatment (including platinum-based chemotherapy. Patients with PD-L1 positivity, TMB-H, or MSI-H/dMMR should have received PD-1/PD-L1 therapy).
     8. Hepatocellular carcinoma: Progression or recurrence after at least second-line treatment.
     9. Renal cell carcinoma: Progression or recurrence after at least second-line treatment.

        Phase IIa:

        The tumor types and biomarker requirements for each expansion cohort in Phase IIa will be further determined based on data from Phase Ib and discussions with the Study Monitoring Committee (SMC).

        4. ECOG performance status ≤1. 5. Life expectancy of ≥12 weeks. 6. Organ function levels must meet the following criteria:

     <!-- -->

     1. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
     2. Hemoglobin (HGB) ≥90 g/L;
     3. Platelet count (PLT) ≥100×10^9/L;
     4. Serum creatinine ≤1.5×ULN or estimated creatinine clearance ≥60 mL/min (according to the Cockcroft and Gault formula);
     5. Serum total bilirubin (TBil) ≤1.5×ULN. For participants with liver metastases or Gilbert's syndrome, TBil >1.5×ULN is allowed if direct bilirubin (DBil) is <ULN. AST and ALT ≤2.5×ULN. For participants with liver metastases or Gilbert's syndrome, AST/ALT ≤5×ULN is allowed.

        7. Willingness to participate in this study and provision of informed consent. 8. All acute toxicities from previous anticancer treatments or surgical procedures must have resolved to baseline severity or to NCI-CTCAE Version 5.0 ≤Grade 1 (except for alopecia or other toxicities deemed by the investigator to pose no safety risk to the participant).

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for the trial:

1. Known severe allergy to the investigational drug, any of the combination drugs, or any of their excipients (hydroxypropyl-beta-cyclodextrin, arginine, tromethamine, mannitol).
2. Presence or history of other malignancies (except adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, or cervical carcinoma in situ), unless the participant has undergone curative treatment and has evidence of no recurrence or metastasis within the past 5 years.
3. Symptomatic central nervous system (CNS) metastases or CNS metastases requiring corticosteroid treatment within 2 weeks before the first dose of the study drug. Participants with asymptomatic CNS metastases are also excluded. Participants with leptomeningeal carcinomatosis or meningeal dissemination are excluded.
4. Participants with a history of anti-tumor treatment meeting the following criteria must be excluded:

   1. Received mitomycin C or nitrosourea chemotherapy (e.g., carmustine, lomustine) within 6 weeks before the first dose.
   2. Received systemic anti-tumor treatment (e.g., chemotherapy, endocrine therapy, immunotherapy, biological therapy) within 4 weeks before the first dose.
   3. Received investigational drug treatment in a clinical trial or is currently participating in another clinical trial within 4 weeks before the first dose.
   4. Received oral fluoropyrimidine or small-molecule targeted therapy within 2 weeks before the first dose or within 5 half-lives of the known drug (whichever is longer).
   5. Received palliative local radiotherapy within 2 weeks before the first dose.
   6. Received traditional Chinese medicine or patent Chinese medicine with anti-tumor indications within 2 weeks before the first dose.

   Note: If a participant has received multiple treatments with different washout periods, the actual washout period will be determined by the longer duration.
5. Participants who have previously received HDAC inhibitors.
6. Participants who have previously received any estrogen receptor degraders, including but not limited to fulvestrant, are not eligible for the cohort combining with fulvestrant.
7. Participants who have previously received anti-PD-1/PD-L1 antibody treatment are not eligible for the cohort combining with tislelizumab, unless the participant has previously benefited from anti-PD-1/PD-L1 treatment in the advanced/metastatic setting and may be included.
8. Participants with a severe infection within 4 weeks before the first dose of PM (Purinostat Mesylate), or those with active infections requiring oral or intravenous antibiotic treatment within the last 2 weeks.
9. Participants who received transfusions, recombinant human thrombopoietin, recombinant human interleukin-11, erythropoiesis-stimulating agents, or granulocyte colony-stimulating factors within 2 weeks before the first dose of the study drug.
10. For breast cancer: Participants with symptomatic, visceral metastatic disease at high risk of life-threatening complications in the short term (patients with visceral crisis) or inflammatory breast cancer.
11. Participants who experienced ≥Grade 3 immune-related adverse events during previous immunotherapy are not eligible for the cohort combining with tislelizumab.
12. Participants with active or a history of autoimmune diseases that are at risk of recurrence (e.g., systemic lupus erythematosus, rheumatoid arthritis, vasculitis) are not eligible for the cohort combining with tislelizumab. Exceptions include participants with Type I diabetes or autoimmune thyroiditis that can be managed with replacement therapy.
13. Participants who received systemic corticosteroids (prednisone >10 mg/day or equivalent) or other immunosuppressive agents within 14 days before the first dose of PM are not eligible for the cohort combining with tislelizumab.

    Exceptions include the use of topical, ocular, intra-articular, nasal, and inhaled corticosteroids, and short-term corticosteroids for prophylactic treatment (e.g., prior to contrast administration).
14. Participants with uncontrolled or significant cardiovascular or cerebrovascular diseases, including:

    1. New York Heart Association (NYHA) Class II or higher congestive heart failure, unstable angina, myocardial infarction within 6 months before the first dose of PM, or arrhythmias requiring treatment, left ventricular ejection fraction (LVEF) <50% at screening.
    2. Primary cardiomyopathies (e.g., dilated, hypertrophic, arrhythmogenic right ventricular, restrictive, or unclassified cardiomyopathy).
    3. Symptomatic coronary artery disease requiring pharmacological treatment during the screening period.
    4. History of clinically significant QTcF interval prolongation, or an average corrected QT interval (QTc) >450 msec (male) or >470 msec (female) based on three electrocardiograms (ECGs) during screening (repeat and average three values only if the first ECG shows QTc >450 msec (male) or >470 msec (female)); history of long QT syndrome or confirmed family history of long QT syndrome; history of clinically significant ventricular arrhythmias, or current use of antiarrhythmic drugs or implantable defibrillators for ventricular arrhythmias.
    5. Cerebrovascular accident (including intracerebral hemorrhage, cerebral infarction, transient ischemic attack) within 6 months before the first dose of PM.
    6. Inadequately controlled blood pressure during the screening period (regardless of whether antihypertensive medication is being taken): systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg.
    7. Other cardiovascular or cerebrovascular diseases deemed by the investigator as unsuitable for enrollment.
15. Uncontrolled electrolyte disturbances that may affect the action of QTc-prolonging drugs (e.g., hypocalcemia <1.0 mmol/L, hypokalemia <lower limit of normal, hypomagnesemia <0.5 mmol/L), but retesting is allowed after intervention.
16. Current or history of any severity of interstitial lung disease with significant impairment of pulmonary function.
17. Presence of third-space effusions (e.g., pleural effusion, ascites) that cannot be controlled by drainage or other methods.
18. Participants who underwent major surgery requiring general anesthesia within 4 weeks before the first dose of PM or have not withdrawn from other clinical trials; those who underwent surgery requiring local anesthesia/epidural anesthesia within 2 weeks before enrollment and have not recovered (except for tissue biopsy).
19. Clinically significant active infections, including hepatitis B (HBV) and hepatitis C (HCV). Active hepatitis B is defined as participants who are HBsAg positive or HBcAb positive with HBV-DNA above the limit of detection (i.e., upper limit of normal for the laboratory of each center). If participants achieve HBV-DNA negativity after antiviral therapy and are willing to continue antiviral therapy during the study, they may be enrolled after receiving at least 2 weeks of antiviral treatment before the first dose. Active hepatitis C is defined as HCV antibody positive with HCV-RNA above the limit of detection (upper limit of normal). Positive Treponema pallidum antibody (TPAb) and positive non-treponemal antibody titer.
20. History of immunodeficiency, including positive HIV antibody test, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.
21. Participation in another interventional clinical trial within 4 weeks before enrollment.
22. Pregnant or breastfeeding women, or those who cannot ensure the use of contraception during the study and for at least 6 months after the last dose of Purinostat.
23. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk of participation in the study or the risk associated with the administration of the study drug, or may interfere with the study results, as well as other situations where the investigator deems the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | Up to week 96
  defined as the proportion of subjects with an overall efficacy response of complete remission (CR) or partial remission (PR) after at least one post-baseline evaluation during the trial.

SECONDARY OUTCOMES:
Complete Remission Rate (CRR) | Up to week 96
  defined as the proportion of subjects with an overall efficacy response of CR after at least one post-baseline evaluation during the trial;
Disease Control Rate (DCR) | Up to week 96
  defined as the proportion of subjects with an overall efficacy response of CR, PR and stable disease (SD) after at least one post-baseline evaluation during the trial;
Duration of remission (DOR) | Up to week 96
  defined as the duration from first remission (PR and CR) to disease progression or death;
Time to Tumor Remission (TTR) | Up to week 96
  defined as the time from first dose to the appearance of PR or CR;
Progression-free survival (PFS) | Up to week 96
  defined as the time from first dose to disease progression or death
Overall survival (OS) | Up to week 96
  defined as the time from first dose to death.

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Yongsheng Wang, Doctor, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guanzhou, Guangzhou
  - West China hospital of Sichuan university, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No